CLINICAL TRIAL: NCT07125625
Title: Randomized Double Blind Placebo Controlled Trial on a Probiotic Mixture (L. Rhamnosus GG Plus L. Plantarum 299V) in Pediatric Irritable Bowel Syndrome: Clinical Efficacy and Multiomics Approach
Brief Title: Probiotic Mixture (L. Rhamnosus GG and L. Plantarum 299V) In Pediatric Irritable Bowel Syndrome
Acronym: PRIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRIME
Record Dates: First submitted 2025-06-26; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: food supplement; probiotics; irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized double bind with placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Nobody knows the randomization code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 62 children will take the product under study based on One capsule/sachet containing L. Rhamnosus GG 1x10^10 CFU plus L. Plantarum 299V 1x10^10 CFU per day for 8 weeks
  Interventions: Dietary Supplement: Experimental arm: probiotic
- Placebo (Placebo Comparator): 62 children will take a carbohydrate-based control product (maltodextrin)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental arm: probiotic — a dietary supplement containing L. Rhamnosus GG 1x1010 CFU plus L. Plantarum 299V. 1x1010 CFU
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo (maltodextrine)
  Arms: Placebo

SUMMARY:
What is this study about? This clinical study aims to investigate whether a specific combination of probiotics-Lactobacillus rhamnosus GG and Lactobacillus plantarum 299V-can help children and adolescents with Irritable Bowel Syndrome (IBS). IBS is a common digestive condition in children, causing abdominal pain, bloating, and changes in bowel habits (either diarrhoea, constipation, or alternating between the two). These symptoms can seriously affect a child's daily life and wellbeing.

The study is coordinated by the University of Bari, in collaboration with the University of Udine, and led by Prof. Ruggiero Francavilla.

Why is this study being done? Although probiotics are increasingly used in IBS, solid scientific evidence in children is still limited. This study will assess whether the chosen probiotic mix improves symptoms, bowel habits, and quality of life in young people with IBS. It will also investigate how the probiotics affect gut bacteria (microbiota) and the chemicals produced by the body (metabolomics), to better understand how these changes might help relieve symptoms.

Who can take part? Children and adolescents aged 4 to 18 years with a diagnosis of IBS (based on international Rome IV criteria) who experience abdominal pain on a daily basis.

Children with other significant medical conditions, recent surgery, or ongoing infections, as well as those taking antibiotics or other probiotics shortly before the study, cannot participate.

How does the study work? The study is a randomised, double-blind, placebo-controlled trial, meaning that some children will receive the probiotic drops, and others will receive placebo drops (which do not contain probiotics), and neither the participants nor the doctors will know who is receiving which treatment. This is the best way to test whether the probiotics really work.

Each participant will be involved in the study for about 14 weeks, divided into:

A 2-week "run-in" period to confirm eligibility.

An 8-week treatment period (probiotic or placebo).

A 4-week follow-up.

The probiotics/placebo are taken as 20 drops once daily for 8 weeks.

Throughout the study, children and parents will be asked to keep a daily diary of abdominal pain and bowel habits, and to complete validated questionnaires on symptom severity and quality of life. Stool and urine samples will also be collected at different time points to analyse changes in gut bacteria and body metabolism.

What are the aims of the study?

Primary aim:

To see whether the probiotics reduce abdominal pain by at least 30% compared to the start of the study.

Secondary aims:

To check if bowel habits improve (stool consistency and frequency).

To assess improvements in quality of life.

To analyse whether the probiotics cause positive changes in gut bacteria and metabolic profiles.

To ensure that the treatment is safe and well-tolerated.

What are the possible risks and benefits? The probiotic mixture used in this study has been studied in children before and is generally considered safe. The study includes careful monitoring for any side effects.

Participants may or may not experience an improvement in symptoms. However, the information gained from the study will help doctors better understand how probiotics work in IBS and may benefit future patients.

What are participants' rights? Participation is voluntary, and families may withdraw their child from the study at any time, without affecting the child's medical care. The study has been approved by an independent ethics committee and complies with all European and Italian regulations regarding research in children.

All personal data and medical information will be treated confidentially and securely, in accordance with privacy laws.

Where is the study taking place? The study is being conducted at the Paediatric Gastroenterology Unit of the University of Bari Aldo Moro and the Paediatric Unit of the University of Udine. These centres are national referral centres for children with gastrointestinal problems.

Who is funding and organising the study? The study is sponsored and conducted by the University of Bari. The probiotic and placebo products are provided by Dicofarm S.p.A., who also ensures that the placebo and probiotic products look and taste the same to maintain the study's blinding.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is one of the most prevalent functional gastrointestinal disorders in children and adolescents, with an estimated global prevalence ranging from 6% to 14% depending on diagnostic criteria used. IBS is characterized by chronic abdominal pain and altered bowel habits, including diarrhea, constipation, or mixed patterns, in the absence of identifiable structural or biochemical abnormalities. These symptoms significantly impair the quality of life, school performance, and psychosocial well-being of affected individuals.

The pathophysiology of IBS remains multifactorial and incompletely understood. Emerging evidence suggests that disturbances in the gut-brain axis play a critical role, with bidirectional signaling pathways involving the enteric nervous system, central nervous system, and endocrine components. Additionally, alterations in the intestinal microbiota-commonly termed dysbiosis-have been implicated as potential contributors to IBS pathogenesis. Reduced microbial diversity and imbalances in beneficial versus pathogenic bacterial populations have been observed in pediatric IBS patients. Concurrently, immune dysregulation with low-grade mucosal inflammation and altered immune responses may exacerbate symptoms.

The use of probiotics has emerged as a promising therapeutic strategy for managing IBS.

In this context, Lactobacillus rhamnosus GG is one of the most extensively studied probiotics, demonstrating efficacy in improving abdominal pain, stool consistency, and microbial composition in pediatric IBS. Similarly, Lactobacillus plantarum 299V has been associated with a reduction in bloating, improvement in stool frequency, and normalization of gut microbiota in adults.

Despite promising preliminary results, robust, high-quality evidence supporting the efficacy of thiscombination in pediatric IBS remains limited, highlighting the need for further investigation.

To address this a large double blind randomized clinical trial including advanced analytical techniques, such as fecal microbiota profiling via 16S rRNA sequencing and urinary metabolomic analysis, provide a unique opportunity to explore the mechanistic underpinnings of probiotic action. Microbiota profiling allows for the identification of specific bacterial taxa changes associated with symptom improvement, while metabolomics can reveal alterations in gut microbial metabolites, such as short chain fatty acids (SCFAs), that may mediate therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-18 years;
* Irritable Bowel Syndrome according to Rome IV criteria
* Average daily pain rate of at least 3 out of 10 VAS met during run-in period •-Written informed consent of parent's/legal tutor and verbal or written assent of the patient based on the minor's maturity

Exclusion Criteria:

* Presence of other gastrointestinal diseases (inflammatory bowel disease, pancreatitis, chronic liver disease, eosinophilic esophagitis, peptic ulcer disease, celiac disease, pseudo-obstruction, small bowel bacterial overgrowth, or Hirschsprung's disease);
* Significant chronic health condition requiring specialty care (e.g., lithiasis, ureteropelvic junction obstruction, sickle cell, cerebral palsy, hepatic, hematopoietic, renal, endocrine, or metabolic diseases) that could potentially impact the child's ability to participate or confound the results of the study.
* Primary or secondary immunodeficiency;
* Malnutrition;
* History of abdominal surgery in the past 3 months.;
* Chronic or acute infectious diseases (viral, bacterial, parasitic) in progress;
* Rome IV criteria diagnosis of functional constipation.
* Use of probiotics/antibiotics within 4 weeks prior to enrolment;
* Current pregnancy or breastfeeding;
* Psychiatric conditions that reduce compliance with the protocol.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
VAS visual analogue scale 0-10 | BASELINE AND AFTER 4 WEEKS
  Treatment success defined as decrease of abdominal pain severity of at least 30% from baseline (measured with VAS).

SECONDARY OUTCOMES:
Bristol Stool Form Scale | BASELINE AND AFTER 4 WEEKS
  Stool consistency improvement measured with Bristol Stool Form Scale (≥1 Bristol Stool Form Scale to a higher number average consistency at the last week of trial compared with baseline for IBS-D or lower number for IBS-C) between baseline and end of treatment in the two groups
Change in Quality of life | BASELINE AND AFTER 4 WEEKS
  Change in Quality of life as assed by Pediatric Quality of Life Inventory 4.0 between baseline and end of treatment in the two groups
Irritable Bowel Syndrome Symptom Severity Score | BASELINE AND AFTER 4 WEEKS
  Change in IBS severity as measured by the Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) between baseline and end of treatment in the two groups
Microbiota | BASELINE AND AFTER 4 WEEKS
  Changes in the microbiota composition as well as changes in the fecal and urinary metabolomic profiles between baseline and end of treatment in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatria Trambusti, Bari, bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Varni JW, Limbers CA, Burwinkle TM. How young can children reliably and validly self-report their health-related quality of life?: an analysis of 8,591 children across age subgroups with the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jan 3;5:1. doi: 10.1186/1477-7525-5-1. PMID 17201920
- [Background] Varni JW, Lane MM, Burwinkle TM, Fontaine EN, Youssef NN, Schwimmer JB, Pardee PE, Pohl JF, Easley DJ. Health-related quality of life in pediatric patients with irritable bowel syndrome: a comparative analysis. J Dev Behav Pediatr. 2006 Dec;27(6):451-8. doi: 10.1097/00004703-200612000-00001. PMID 17164617
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Self MM, Czyzewski DI, Chumpitazi BP, Weidler EM, Shulman RJ. Subtypes of irritable bowel syndrome in children and adolescents. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1468-73. doi: 10.1016/j.cgh.2014.01.031. Epub 2014 Jan 29. PMID 24486406
- [Background] Lane MM, Czyzewski DI, Chumpitazi BP, Shulman RJ. Reliability and validity of a modified Bristol Stool Form Scale for children. J Pediatr. 2011 Sep;159(3):437-441.e1. doi: 10.1016/j.jpeds.2011.03.002. Epub 2011 Apr 13. PMID 21489557
- [Background] Chumpitazi BP, Lane MM, Czyzewski DI, Weidler EM, Swank PR, Shulman RJ. Creation and initial evaluation of a Stool Form Scale for children. J Pediatr. 2010 Oct;157(4):594-7. doi: 10.1016/j.jpeds.2010.04.040. Epub 2010 Jun 17. PMID 20826285
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] Korpela K, Salonen A, Virta LJ, Kekkonen RA, Forslund K, Bork P, de Vos WM. Intestinal microbiome is related to lifetime antibiotic use in Finnish pre-school children. Nat Commun. 2016 Jan 26;7:10410. doi: 10.1038/ncomms10410. PMID 26811868
- [Background] Francavilla R, Miniello V, Magista AM, De Canio A, Bucci N, Gagliardi F, Lionetti E, Castellaneta S, Polimeno L, Peccarisi L, Indrio F, Cavallo L. A randomized controlled trial of Lactobacillus GG in children with functional abdominal pain. Pediatrics. 2010 Dec;126(6):e1445-52. doi: 10.1542/peds.2010-0467. Epub 2010 Nov 15. PMID 21078735
- [Background] Trivic I, Niseteo T, Jadresin O, Hojsak I. Use of probiotics in the treatment of functional abdominal pain in children-systematic review and meta-analysis. Eur J Pediatr. 2021 Feb;180(2):339-351. doi: 10.1007/s00431-020-03809-y. Epub 2020 Sep 17. PMID 32940743
- [Background] Saulnier DM, Riehle K, Mistretta TA, Diaz MA, Mandal D, Raza S, Weidler EM, Qin X, Coarfa C, Milosavljevic A, Petrosino JF, Highlander S, Gibbs R, Lynch SV, Shulman RJ, Versalovic J. Gastrointestinal microbiome signatures of pediatric patients with irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1782-91. doi: 10.1053/j.gastro.2011.06.072. Epub 2011 Jul 8. PMID 21741921
- [Background] Tap J, Derrien M, Tornblom H, Brazeilles R, Cools-Portier S, Dore J, Storsrud S, Le Neve B, Ohman L, Simren M. Identification of an Intestinal Microbiota Signature Associated With Severity of Irritable Bowel Syndrome. Gastroenterology. 2017 Jan;152(1):111-123.e8. doi: 10.1053/j.gastro.2016.09.049. Epub 2016 Oct 7. PMID 27725146
- [Background] Collins SM, Surette M, Bercik P. The interplay between the intestinal microbiota and the brain. Nat Rev Microbiol. 2012 Nov;10(11):735-42. doi: 10.1038/nrmicro2876. Epub 2012 Sep 24. PMID 23000955
- [Background] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632